CLINICAL TRIAL: NCT00492076
Title: A Randomised, Double-Blind Placebo-Controlled Study Assessing the Short-Term Effect of a Dermatophagoides Pteronyssinus Extract, Quantified in Mass Units, in Subjects With Perennial Mite Induced Asthma
Brief Title: Efficacy and Safety Trial of Subcutaneous Immunotherapy in Mite Induced Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Fernando de la Torre/medical marketing manager, ALK-ABELLO, S.A.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: E04/05/PP-M
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Allergic Asthma
Keywords: Specific immunotherapy; Mite; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Pangramin Plus Dermatophagoides pteronyssinus 100%
  Interventions: Biological: Pangramin Plus D. pteronyssinus 100%
- 2 (Placebo Comparator): Pangramin Plus placebo
  Interventions: Biological: Pangramin Plus D. pteronyssinus 100%

INTERVENTIONS:
Biological: Pangramin Plus D. pteronyssinus 100% — 1. Active. Pangramin Plus D. pteronyssinus 100%
  2. Placebo. Pangramin Plus placebo

SUMMARY:
The purpose of this study is to determine whether a short course of subcutaneous immunotherapy is efficacious in mite induced asthma. The efficacy is based on reduction in control medication.

DETAILED DESCRIPTION:
The control of mild-moderate persistent asthma include the need of concomitant medication, as inhaled corticosteroids. However, compliance in perennial asthma is low. The aim of this study is to assess the possibility to reduce the need of concomitant medication through a short-course of subcutaneous immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Mild/moderate persistent asthma
* Positive skin prick test or specific IgE to mites
* Age: 14-55 years old

Exclusion Criteria:

* Immunotherapy contraindications
* Allergy to other inhalant allergens
* Previous immunotherapy (5 years)with mites

Ages: 14 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Reduction in inhaled corticosteroids | 4 months

SECONDARY OUTCOMES:
Reduction in symptoms and rescue medication Tolerability | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ana I Tabar, MD PhD, Principal Investigator — Hospital Virgen del Camino
Locations (1):
- Hospital Virgen del Camino, Allergology Service, Pamplona, Navarre, Spain